CLINICAL TRIAL: NCT03118154
Title: Efficacy of Manual Therapy to Improve Quality of Life and Decrease Pain in Subjects With Endometriosis
Acronym: Endo2017
Status: Terminated | Type: Observational
Why Stopped: Recruitment
Sponsor: Clear Passage Therapies, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: ENDO-2017-C0100
Record Dates: First submitted 2017-04-05; First posted 2017-04-18 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Endometriosis; Pelvic Pain; Dysmenorrhea
Keywords: endometriosis; pelvic pain; dysmenorrhea
MeSH Terms: conditions — Endometriosis; Pelvic Pain; Dysmenorrhea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Manual Physical Therapy, retrospective: Endometriosis subjects treated at Clear Passage with follow up to assess changes in pain and overall health in a retrospective chart review.
  Interventions: Other: Manual Physical Therapy
- Control, prospective: Endometriosis control subjects not treated at Clear Passage that complete two questionnaires, 30 days apart, to assess changes in their pain levels.

INTERVENTIONS:
Other: Manual Physical Therapy — Manual Physical Therapy intervention using the Clear Passage Approach (CPA). The focus of the CPA is to deform adhesions throughout the body using a variety of manual therapy techniques and modalities.
  Groups: Manual Physical Therapy, retrospective

SUMMARY:
This study will compare subjects with a history of pelvic or menstrual pain diagnosed with endometriosis treated at Clear Passage with untreated control subjects. The treatment group will be a retrospective chart review; the control subject group will be a prospective questionnaire based study.

The study will assess the changes in pain experienced by subjects treated with manual therapy at Clear Passage to untreated subjects with endometriosis.

DETAILED DESCRIPTION:
This study has two segments the first is a chart and outcome assessment of patients treated at Clear Passage (CP) with a diagnosis of endometriosis. These patients have completed multiple questionnaires as a standard of care for outcome monitoring in the clinic setting, no new data will be collected. The second segment is a prospective observational, online questionnaire based study of female subjects with a diagnosis of endometriosis not treated at CP. Data on the impact of quality of life (QOL) over time of subjects not treated at CP will be assessed using the same questionnaire used as standard of care in the clinic twice, 30 days apart. This will be accomplished using online forms with subjects able to complete the questionnaires with ease via the internet. The data obtained from the untreated subjects will allow for reporting of overall impact on QOL in this population, as well as provide a control group for assessment of improvement for manual therapy interventions for patients with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of endometriosis
* Experience either pain with menstruation or other pelvic pain
* Able to complete the questionnaires online

Exclusion Criteria:

* Currently pregnant
* Cancer diagnosis
* Prior chemotherapy or radiation treatment(s)
* Prior treatment at Clear Passage

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study focuses on female subjects with a medical diagnosis of endometriosis that experience pain with menstruation or pelvic pain not associated with menstruation between the ages of 18 and 65.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2017-10-01 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
Reported overall pain rating | 30 days
  Self reported values using the Pain Questionnaire
Reported Global Health | 30 days
  Self reported values using the Global Health Questionnaire
Reported Pain Intensity | 30 days
  Self reported values using the Pain Interference Questionnaire
Reported Sexual Function | 30 days
  Self reported values using the Female Sexual Function Index Questionnaire

SECONDARY OUTCOMES:
Correlations to positive treatment outcomes | 30 days
  Medical history correlations for positive outcomes in subjects treated with manual therapy

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence J Wurn, LMT, Principal Investigator — Clear Passage Therapies
Locations (1):
- Clear Passage Physical Therapy, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rice AD, Patterson K, Wurn BF, King CR and Wurn LJ. Update on "Decreasing dyspareunia and dysmenorrhea in women with endometriosis via a manual physical therapy: results from 2 independent studies". Journal of Endometriosis and Pelvic Pain Disorders, 6(3):161-162, 2014.
- [Background] Wurn BF, Wurn LJ, Patterson K, King CR, Scharf ES. Decreasing dyspareunia and dysmenorrhea in women with endometriosis via a manual physical therapy: Results from two independent studies. Journal of Endometriosis and Pelvic Pain Disorders 3(4):188-196, 2011.